CLINICAL TRIAL: NCT05266599
Title: The Effect of Two Different Root Canal Sealers on Postobturation Pain in Single-Visit Root Canal Treatment: A Prospective Clinical Randomized Study- Part 1, Influence of Resin-based and Mineral Trioxide Aggregate-based Sealers on Treatment Outcome After Two-year Follow-up in Mandibular Molar Teeth With Asymptomatic Irreversible Pulpitis-Part 2
Brief Title: The Effect of Two Different Root Canal Sealers on Postobturation Pain and Clinical and Radiographical Outcome After Two-year Follow-up
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ege University (Other)
Responsible Party: Principal Investigator, Gözde Kandemir Demirci, Principal Investigator, Ege University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 19-11/6
Record Dates: First submitted 2022-02-19; First posted 2022-03-04 (Actual); Last update posted 2022-03-04 (Actual); Status verified 2022-03

CONDITIONS: Asymptomatic Vital Mandibular Molar Teeth
Keywords: asymptomatic irreversible pulpitis; bioceramic sealer; post-obturation pain; resin-based sealer; treatment outcome
MeSH Terms: interventions — epoxy resin-based root canal sealer

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MTA Fillapex group (Active Comparator): Root canals were prepared with WaveOne Gold instruments and X-Smart Plus (Dentsply Maillefer, Switzerland) endodontic motor. Final irrigation was performed with 5 ml of 17% ethylene diamine tetraacetic acid (EDTA), 5 ml of 2.5% NaOCl, and distilled water. Then, the root canals were dried with the help of sterilized paper cones. MTA Fillapex sealer was mixed and applied to the root canals and the main gutta-percha cone. Then, the single cone technique was utilized for the obturation of the root canals.
  Interventions: Other: MTA Fillapex root canal sealer
- AH Plus group (Active Comparator): Root canals were prepared with WaveOne Gold instruments and X-Smart Plus (Dentsply Maillefer, Switzerland) endodontic motor. Final irrigation was performed with 5 ml of 17% ethylene diamine tetraacetic acid (EDTA), 5 ml of 2.5% NaOCl, and distilled water. Then, the root canals were dried with the help of sterilized paper cones. AH Plus sealer was mixed and applied to the root canals and the main gutta-percha cone. Then, the single cone technique was utilized for the obturation of the root canals.
  Interventions: Other: AH Plus root canal sealer

INTERVENTIONS:
Other: MTA Fillapex root canal sealer — Root canal treatments were performed with MTA Fillapex
  Arms: MTA Fillapex group
Other: AH Plus root canal sealer — Root canal treatments were performed with AH plus
  Arms: AH Plus group

SUMMARY:
Post-obturation pain evaluation(Part 1):

One hundred asymptomatic mandibular molar teeth with vital pulp were randomly assigned into two groups according to the sealer used MTA Fillapex (Angelus Odontologica Industries SA, Londrina, PR, Brazil) or AH Plus (Dentsply Sirona, Ballaigues, Switzerland) sealer. WaveOne Gold instruments were used for root canal preparations in both groups. Root canals were obturated with the manufacturer advised own gutta-percha points of preparation technique and MTA Fillapex was used in the first group and AH Plus was used in the second group as a root canal sealer. Postoperative pain at 6, 12, 24, 48, 72 hours, 4, 5, 6, 7, and 30 days after root canal treatment was measured with the Numerical Rating Scale (NRS), and patients were informed to record the number of analgesics they used during these time periods.

Clinical and radiological outcome evaluation(Part 2):

Patients were recalled for clinical and radiographic examinations at 12 and 24 months postoperatively. The clinical outcome was determined as success or failure according to objective evaluation of symptoms of inflammation or infection. In clinical examination at follow-up appointments, swelling, pain, sinus tract, tenderness to percussion, and/or palpation test, periodontal probing depths were determined and recorded. The radiographic outcome was evaluated and classified according to the Strindberg criteria. Teeth with a normal contour, width, and structure of the periodontal ligament were considered as"successful" and teeth with a widened periodontal contours or a new periapical radiolucency were considered as "failed". Additionally, the other parameters (age, gender, tooth number, apical gutta level) on treatment success were examined.

DETAILED DESCRIPTION:
This randomized clinical trial aimed to evaluate and compare the effect of MTA-based bioceramic and resin-based sealers on the incidence and intensity of post-obturation pain and clinical and radiological outcome after two-year follow-up in asymptomatic vital molar teeth in single-visit root canal treatment. One hundred asymptomatic mandibular molar teeth with vital pulp were randomly assigned into two groups according to the sealer used MTA Fillapex (Angelus Odontologica Industries SA, Londrina, PR, Brazil) or AH Plus (Dentsply Sirona, Ballaigues, Switzerland) sealer. WaveOne Gold instruments were used for root canal preparations in both groups. Root canals were obturated with the manufacturer advised own gutta-percha points of preparation technique and MTA Fillapex was used in the first group and AH Plus was used in the second group as a root canal sealer.

Post-obturation pain evaluation(Part 1):

Postoperative pain at 6, 12, 24, 48, 72 hours, 4, 5, 6, 7, and 30 days after root canal treatment was measured with the Numerical Rating Scale, and patients were informed to record the number of analgesics they used during these time periods. The Mann-Whitney U test was used to compare the postoperative pain and the analgesic use between the two groups according to NRS scores. The relationship between the number of analgesics used and the total NRS values were analyzed by Spearman Correlation Analysis. Evaluation of NRS scores at all time points for each group was done by Friedman Two-Way Analysis of Variance Test.

Clinical and radiological outcome evaluation(Part 2):

Patients were recalled for clinical and radiographic examinations at 12 and 24 months postoperatively. The clinical outcome was determined as success or failure according to objective evaluation of symptoms of inflammation or infection. In clinical examination at follow-up appointments, swelling, pain, sinus tract, tenderness to percussion, and/or palpation test, periodontal probing depths were determined and recorded. The radiographic outcome was evaluated and classified according to the Strindberg criteria. Teeth with a normal contour, width, and structure of the periodontal ligament were considered as "successful" and teeth with a widened periodontal contours or a new periapical radiolucency were considered as"failed". Additionally, the other parameters (age, gender, tooth number, apical gutta level) on treatment success were examined. All of the pairwise comparisons between the groups at 1st and 2nd year were done by chi-square test (Fisher exact test). Pearson's chi-square test was used to evaluate the age, gender of the patients and tooth types between the groups

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years
* Good oral hygiene
* Patients with mature mandibular first or second molars diagnosed with asymptomatic irreversible pulpitis due to deep caries
* Teeth that have not been treated endodontically and restoratively before
* A delayed positive response to cold test and electric pulp tests in the vitality test of the teeth
* Large pulpal perforation during caries removal
* Presence of thick and profuse pulpal bleeding could not be controlled within 5 minutes
* Absence of periapical pathology of teeth when confirmed with periapical radiographically

Exclusion Criteria:

* Patients who refused to participate in the study
* The patients are not systemically healthy, allergic to the materials and agents used during root canal treatment
* Having a history of sensitivity to local anesthetics.
* Patients who used antibiotics and analgesics in the 7 days prior to the beginning of treatment.
* Symptomatic or non-vital teeth
* Patients have more than one tooth requiring endodontic treatment
* Teeth with material loss that cannot be restored, or teeth that require a post or that will be used as a supporting tooth for a prosthesis
* The presence of advanced periodontal disease (probing depth >3 mm)
* Presence of calcified root canal, presence of internal or external root resorption
* Second molars with C-shaped root canal anatomy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2019-11-20 (Actual); Primary Completion 2022-02-07 (Actual); Study Completion 2022-02-07 (Actual)

PRIMARY OUTCOMES:
The incidence and intensity of post-obturation pain | up to 30-day
  Post-obturation pain up to 30 days after root canal treatment was measured with Numerical Rating Scale. The Numerical Rating Scale is a pain measurement scale that encompasses the following grades: 0 no pain, 1-3 mild pain, 4-6 moderate pain, 7-10 severe pain.

SECONDARY OUTCOMES:
Clinical and radiographical success with resin-based and MTA-based bioceramic sealer | 1 year and 2 year follow-up
  The clinical outcome was determined as success or failure according to objective evaluation of symptoms of inflammation or infection. In clinical examination, swelling, pain, sinus tract, tenderness to percussion and/or palpation test, periodontal probing depths were determined and recorded. The radiographic outcome was evaluated and classified according to the Strindberg criteria (Strindberg 1956). Teeth with a normal contour, width and structure of the periodontal ligament were considered "successful" and teeth with a widened periodontal contours or a new periapical radiolucency were considered "failed". A case was considered unsuccessful when at least one of the clinical and/or radiographic findings was present. Unsuccessful ones were scored as "0" and successful ones as "1".

CONTACTS AND LOCATIONS:
Overall Officials: Gözde K Demirci, Dr, Principal Investigator — Ege University Faculty of Dentistry; Melis Coşar, Study Chair — Ege University Faculty of Dentistry; Mehmet Kemal Çalışkan, Prof.Dr, Study Chair — Ege University Faculty of Dentistry
Locations (1):
- Gözde Kandemir Demirci, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zavattini A, Knight A, Foschi F, Mannocci F. Outcome of Root Canal Treatments Using a New Calcium Silicate Root Canal Sealer: A Non-Randomized Clinical Trial. J Clin Med. 2020 Mar 13;9(3):782. doi: 10.3390/jcm9030782. PMID 32183124
- [Result] Atav Ates A, Dumani A, Yoldas O, Unal I. Post-obturation pain following the use of carrier-based system with AH Plus or iRoot SP sealers: a randomized controlled clinical trial. Clin Oral Investig. 2019 Jul;23(7):3053-3061. doi: 10.1007/s00784-018-2721-6. Epub 2018 Nov 5. PMID 30397735
- [Result] Aslan T, Donmez Ozkan H. The effect of two calcium silicate-based and one epoxy resin-based root canal sealer on postoperative pain: a randomized controlled trial. Int Endod J. 2021 Feb;54(2):190-197. doi: 10.1111/iej.13411. Epub 2020 Oct 17. PMID 32929721
- [Result] Fonseca B, Coelho MS, Bueno CEDS, Fontana CE, Martin AS, Rocha DGP. Assessment of Extrusion and Postoperative Pain of a Bioceramic and Resin-Based Root Canal Sealer. Eur J Dent. 2019 Jul;13(3):343-348. doi: 10.1055/s-0039-3399457. Epub 2019 Dec 3. PMID 31794999
- [Result] Chybowski EA, Glickman GN, Patel Y, Fleury A, Solomon E, He J. Clinical Outcome of Non-Surgical Root Canal Treatment Using a Single-cone Technique with Endosequence Bioceramic Sealer: A Retrospective Analysis. J Endod. 2018 Jun;44(6):941-945. doi: 10.1016/j.joen.2018.02.019. Epub 2018 Mar 29. PMID 29606401
- [Result] Galani M, Tewari S, Sangwan P, Mittal S, Kumar V, Duhan J. Comparative Evaluation of Postoperative Pain and Success Rate after Pulpotomy and Root Canal Treatment in Cariously Exposed Mature Permanent Molars: A Randomized Controlled Trial. J Endod. 2017 Dec;43(12):1953-1962. doi: 10.1016/j.joen.2017.08.007. Epub 2017 Oct 20. PMID 29061359